CLINICAL TRIAL: NCT05104788
Title: A Phase II, Single-Arm, Prospective Study of Neoadjuvant Icotinib With Chemotherapy for the Treatment of Patients With Epidermal Growth Factor Receptor Mutation Positive, Resectable for Stage II to IIIB(N2) Non-small Cell Lung Cancer
Brief Title: A Study of Icotinib With Chemotherapy as Neoadjuvant Therapy for Patients With EGFRm Positive Resectable Non-Small Cell Lung Cancer
Acronym: NeoIpower
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Wu Nan, Principal Investigator, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV102
Record Dates: First submitted 2021-10-26; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Resectable; NSCLC; Icotinib; EGFRm Positive; Neoadjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icotinib with platinum-based chemotherapy (Experimental): Icotinib 125 mg TID plus investigator's choice of platinum-based standard of care chemotherapy (pemetrexed/carboplatin or pemetrexed/cisplatin)
  Interventions: Drug: Icotinib; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Icotinib — Oral
Drug: Cisplatin — Cisplatin (75mg/m2) to be administered with pemetrexed on Day 1 of every 3-week cycle for 2 cycles.
Drug: Carboplatin — Carboplatin (AUC5) to be administered with pemetrexed on Day 1 of every 3-week cycle for 2 cycles
Drug: Pemetrexed — Pemetrexed (500 mg/m2) to be administered with cisplatin or carboplatin on Day 1 of every 3-week cycle for 2 cycles

SUMMARY:
This is a Phase II, single-Arm, prospective study of neoadjuvant Icotinib with chemotherapy for the treatment of patients with epidermal growth factor receptor mutation positive, resectable for stage II to IIIB(N2) Non-small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Male or female, at least 18 years of age.
* Histologically or cytologically documented lung adenocarcinoma within 60 days prior to study enrollment.
* Clinical stage IIA/IIB/IIIA/IIIB assessed by EBUS-TBNA or PET(positron emission tomography)/CT can be resected.
* EGFR mutation was detected by Amplification Refractory Mutation System(ARMS) and confirmed to be one of the 2 common EGFR mutations known to be associated with EGFR-TKI （epidermal growth factor receptor tyrosine kinase inhibitors）sensitivity (Ex19del, L858R).
* Presence of at least one accurately measurable lesion, CT showing a maximum diameter of 10mm at baseline (except for lymph nodes with a short axis of 15mm required) and suitable for accurate repeat measurements.
* Eastern Cooperative Oncology Group (ECOG) performance status （PS） of 0 or 1 at enrolment.
* Hematology , liver and kidney function are adequate for neoadjuvant therapy.
* Cardiopulmonary function suitable for surgical treatment (ECG, echocardiography, pulmonary function or blood gas analysis).
* Serum pregnancy test (for females of childbearing potential) negative at screening.Female patients of non-childbearing potential must meet at least 1 of the following criteria:

  ① Achieved postmenopausal status, defined as follows: cessation of regular menses forat least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle- stimulating hormone (FSH)level confirming the postmenopausal state;

  ② Have undergone a documented hysterectomy and/or bilateral oophorectomy;

  ③ Have medically confirmed ovarian failure. All other female patients (including female patients with tubal ligations） are considered to be of childbearing potential.
* Male subjects must be willing to use barrier contraception

Exclusion Criteria:

* Mixed squamous cell carcinoma, large cell carcinoma，small cell lung cancer.
* Prior treatment with any systemic anti-cancer therapy for NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug.
* Pregnant female patients; breastfeeding female patients.
* Current use of (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of Cytochrome P450 3A4(CYP3A4)(at least 3 weeks prior).
* Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension and active bleeding, that the investigator considers to be detrimental to patient participation in the study or to adherence to the protocol. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV) or hepatitis C virus (HCV) (e.g., in case of known HBsAg or HCV antibody positivity), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness.
* Clinically significant cardiovascular disease, that is, active or within 3 months prior to enrollment: cerebral vascular accident/stroke, myocardial infarction, unstable angina,congestive heart failure (New York Heart Association Classification Class ≥ II), second-degree or third-degree Atrioventricular（AV）block (unless paced) or any AV block with PR >220 msec; or ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥ 2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless patient is otherwise healthy such as long-distance runners, etc.), machine-read ECG with QTc(corrected QT interval) >470 msec, or congenital long QT syndrome.
* A history of hypersensitivity to Icotinib with or without active excipients or to drugs of similar chemical structure or class, and uncontrollable nausea and vomiting, chronic gastrointestinal disease, inability to swallow formulated drugs, or having undergone major bowel resection that would interfere with adequate absorption of Icotinib.
* Past medical history of Interstitial lung disease（ ILD）, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* Inadequate bone marrow reserve (a leukocyte count less than 4000 mm3, a platelet count less than 100,000 mm3, and a hemoglobin level less than 10 g/dL); adequate renal function deficiency(not normal serum creatinine and blood urea nitrogen levels, and a creatinine clearance level 60 mg/minute); and an inadequate serum aspartate aminotransferase level more than 2.5 times the upper normal limit (UNL) and a serum alanine aminotransferase level more than 2.5 times the UNL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-10-25 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | From date of randomization to an average of 12 weeks after the first dose
  Defined as ≤10% residual cancer cells in the main tumour, as assessed per central pathology laboratory post-surgery

SECONDARY OUTCOMES:
Pathological complete response (pCR) | From date of randomization to an average of 12 weeks after the first dose
  Defined as absence of any residual cancer cells in the dissected tumour samples, including the main tumour and lymph nodes, assessed post-surgery
Overall Survival (OS) | Up to approximately 5.5 years after the last patient is randomized
  Defined as the time from the date of entry to the date of death from any cause.
Disease free survival (DFS) | From date of randomization up to approximately 42 months after date of resection
  DFS is defined as the time from the date of surgery until the first date of disease recurrence (local or distant) or date of death due to any cause, whichever occurs first.
Objective response rate(ORR) | Baseline (Prior to surgery)
  ORR is defined as the percentage of participants having a complete response or a partial response, measured by RECIST 1.1.
Disease control rate(DCR) | Baseline (Prior to surgery)
  DCR is defined as the percentage of participants having a complete response , a partial response and disease stability measured by RECIST 1.1.
R0 surgical resection rate | Post surgery (within one week)
  the proportion of resection margin without macroscopic or microscopic tumor residue (negative resection margin)
Incidence of Adverse Events | From the time of enrollment to either 28-days after the last dose of last study treatment for patients who do not undergo surgery, or 90-days post-surgery
  AE captured by CYCAE 5.0

OTHER OUTCOMES:
EGFR Mutation Detection of plasma samples for the following-up patients who take TKI. | Up to 8 days
  Monitor the change of plasma EGFR mutation copy number before neoadjuvant therapy, cycle 2 chemotherapy and pre-surgery.
Change Between Pre-treatment and Post-treatment SUVmax (Standardized Uptake Values) in primary tumor and metastatic lymph node. | Up to 8 weeks
  The reduction degree of SUVmax in primary tumor and metastatic lymph nodes before and after neoadjuvant therapy was detected by PET-CT.

CONTACTS AND LOCATIONS:
Locations (1):
- BeijingCancerH, Beijing, China